CLINICAL TRIAL: NCT02358226
Title: HIV & Drug Abuse Prevention for South African Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mary Jane Rotheram-Borus, Director, Global Center for Children and Families, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA038675 (NIH); 1R01DA038675-01A1 (NIH)
Record Dates: First submitted 2014-11-24; First posted 2015-02-06 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Substance-Related Disorders; Human Immunodeficiency Virus; Alcoholism
Keywords: Substance-Related Disorders; Human Immunodeficiency Virus; Alcoholism; South Africa; Men; Soccer; Vocational Training
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Alcoholism; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Soccer League (SL) (Experimental): In the SL arm, participants will be invited to participate in a Soccer League, led by coaches who meet the criteria of: 1) soccer skills, 2) being a role model, and 3) social competence. Coaches will undergo intensive training in ethics; role-playing the delivery of health messages; conducting brief interventions for alcohol; how to acquire information on HIV, TB, alcohol use and employment; linkages to local clinics, data collection; and Street Smart, an evidence-based intervention for high-risk youth. Coaches will provide pre- and post-game talks, incorporating the topics of alcohol and drugs; interacting positively with health care providers, partners and family members; HIV, diabetes; daily routines; healthy social networks; making and saving money; loyalty and national success.
  Interventions: Behavioral: Soccer League (SL)
- Soccer League/Vocational Training (SL-V) (Experimental): The SL-V arm will include both the SL intervention as well as access to Vocational Training through either Silulo Ulutho Technologies, which offers computer courses, or Zenzele Training and Development programs, which provides training in woodwork and wielding. Both programs are located in Khayelitsha, which is close to participants' homes, thus avoiding transport-related barriers. Additionally, the training programs occur in a mentor-mentee context so that participants can develop the interpersonal skills required for employment.
  Interventions: Behavioral: Soccer League/Vocational Training (SL-V)
- Control Condition (CC) (No Intervention): Participants in the CC arm will routinely receive flyers with picture stories regarding HIV prevention strategies and how to access these strategies: HIV testing, circumcision, HIV treatment, including ARV, condoms and sexually transmitted diseases.

INTERVENTIONS:
Behavioral: Soccer League (SL) — Participants will be invited to attend soccer practice in the late afternoons, roughly 2-3 times per week. Competitive games will be held on Saturdays so that friends and family may attend. Using a mobile phone application, coaches will regularly record information on participants' arrival and departure times, sportsmanship, volunteering in the community, the results of saliva tests for drugs and alcohol. The SL intervention arm will last for one year.
  Arms: Soccer League (SL)
Behavioral: Soccer League/Vocational Training (SL-V) — In addition to the SL intervention, participants will gain access to vocational training. The Vocational Training will take place through the Silulo or Zenzele programs based in Khayelitsha for a period of 6 months. These programs offer practical and market-related training in computer skills, woodwork, or welding. The SL-V intervention arm will last for one year; with six months dedicated to soccer and six months dedicated to vocational training.
  Arms: Soccer League/Vocational Training (SL-V)

SUMMARY:
The purpose of this study is to test the efficacy of randomizing all young men in a neighborhood to receive: 1) soccer training; 2) soccer and vocational training; or 3) a control condition, as a means to engage young men in HIV prevention. The investigators hypothesize that the intervention will reduce young men's substance use and increase HIV testing.

DETAILED DESCRIPTION:
South Africa has the highest number of HIV-infected persons of any nation, including 2.4 million men, and from 2002-2011 young men have had a 3% incidence HIV rate that has remained stable. New infections occur later in men than in women, making men in their 20s a target for intervention. Decreasing sexual risk and concurrent partnerships is a key outcome in interventions to reduce HIV incidence. Most men (68%) report unprotected sex, typically with three partners in the last three months,and more than half of young men do not use condoms with casual partners.

In South Africa, the amount of alcohol consumed per adult is among the highest in the world. 'Heavy episodic drinking', which most strongly correlates with risky sexual behaviors and HIV infection, is reported by 60% of men. Alcohol, tik (methamphetamine) and marijuana are common among young men in South Africa. Among alcohol abusers, men are highly likely to be poly substance users. Among HIV seropositive young men, drug use is common. Drug and alcohol use is associated with risky sexual behaviors and an increase in the number of sexual partners.

In townships, alcohol is involved in or responsible for 60% of automobile accidents, 75% of homicides, 50% of non-natural deaths, 67% of domestic violence, 30% of hospital admissions, and costs South Africa about R9 billion annually. Violence also characterizes the lives of young men in the Xhosa townships. Intimate partner violence is frequent in alcohol-using partnerships and is correlated with increased HIV incidence. Substance use and unemployment often lead to violence in a township. Jobs, by contrast, provide income and create a strong and respected community role.

HIV prevention efforts for young people in Sub-Saharan Africa have largely been unsuccessful: novel, structural, community level programs that address the social determinants of HIV are needed. Unemployment and a culture of alcohol and violence are major social determinants of HIV among young men. Yet, men are often excluded from economic development programs. Young, South African men need new pathways for prosocial roles and behaviors and our interventions need to be attractive and consistent with men's styles. The social determinants of HIV (unemployment, alcohol, and violence) are critical to creating opportunities for prosocial roles for young men. One of the most common comments by both the men and their families in our previous pilot qualitative study on soccer and vocational training was men's lack of "things to do." Given these needs, the investigators focus on soccer and vocational training in this randomized controlled trial as opportunities for young men to acquire the habits of daily living that are most likely to result in jobs, health, and positive relationships.

ELIGIBILITY:
Inclusion Criteria:

* not employed
* sleeps at least 4 nights per week in the two months prior to recruitment in a household in the target neighborhood boundaries
* speaks Xhosa or English
* provides voluntary informed consent and understands the consent process
* does not appear to be actively hallucinating or incapable of understanding the interviewer

Exclusion Criteria:

* if the interviewer reports that the young man demonstrates delusional talk or cannot comprehend the voluntary informed consent forms

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1211 (Actual)
Dates: Start 2016-05; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the number of outcomes out of 15 outcomes significantly favoring the intervention over the control (Harwood, Weiss & Comulada, 2017) | Baseline to 18 months
  The primary outcome is the number of 15 outcomes (listed shortly) in which the intervention groups are better at the end of the study at 18 months. The outcomes are documented by biomarkers or self-report and except where otherwise noted, are in reference to the last three months. The outcomes are - (1) no concurrent partnerships; (2) no sex without condoms; (3) employment (part/full-time); (4) income above 1200 ZAR/month; (5) no violent acts toward women; (6) no arrests by police; (7) engaged in a community activity; (8) CES-D score < 16 (i.e., caseness); (9) AUDIT score < 3 (i.e., problematic alcohol use); (10) no alcohol usage in last 24 hours; (11) HIV testing; (12) no marijuana (dagga) usage in the last 10 days; (13) no quaalude (mandrax) usage in the last 2-3 days; (14) no methamphetamine (tik) usage in the last 1-2 days; and, (15) PEth Alcohol Test (excessive alcohol use in prior 3 weeks, at 18 months only).

SECONDARY OUTCOMES:
If a significant number of the 15 outcomes have intervention groups better than control at the end of the study, we will analyze and report on each outcome separately. | Baseline to 18 months
  The outcomes are documented by biomarkers or self-report and except where otherwise noted, are in reference to the last three months. The outcomes are - (1) no concurrent partnerships; (2) no sex without condoms; (3) employment (part/full-time); (4) income above 1200 ZAR/month; (5) no violent acts toward women; (6) no arrests by police; (7) engaged in a community activity; (8) CES-D score < 16 (i.e., caseness); (9) AUDIT score < 3 (i.e., problematic alcohol use); (10) no alcohol usage in last 24 hours; (11) HIV testing; (12) no marijuana (dagga) usage in the last 10 days; (13) no quaalude (mandrax) usage in the last 2-3 days; (14) no methamphetamine (tik) usage in the last 1-2 days; and, (15) PEth Alcohol Test (excessive alcohol use in prior 3 weeks, at 18 months only).
Among HIV+, uptake and adherence to ARV medications and medical regimens | Baseline to 18 months
  Assessed via repeated self-reports over 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Rotheram, PhD, Principal Investigator — Department of Psychiatry & Biobehavioral Sciences, Semel Institute, UCLA
Locations (1):
- Stellenbosch University, Stellenbosch, South Africa

REFERENCES:
- [Background] UNAIDS, WHO, & UNICEF. (2011). Global HIV/AIDS response: epidemic update and health sector progress towards universal access (progress report 2011). Geneva, Switzerland: UNAIDS, WHO, & UNICEF.
- [Background] Barnighausen T, Tanser F, Newell ML. Lack of a decline in HIV incidence in a rural community with high HIV prevalence in South Africa, 2003-2007. AIDS Res Hum Retroviruses. 2009 Apr;25(4):405-9. doi: 10.1089/aid.2008.0211. PMID 19320571
- [Background] Statistics South Africa. (2013). Quarterly Labour Force Survey: Quarter 2, 2013. Cape Town, South Africa: Statistics South Africa.
- [Background] Aral SO, Peterman TA. Measuring outcomes of behavioural interventions for STD/HIV prevention. Int J STD AIDS. 1996;7 Suppl 2:30-8. doi: 10.1258/0956462961917753. No abstract available. PMID 8799792
- [Background] Epstein, H. (2007). The invisible cure: Africa, the West, and the fight against AIDS. New York, NY: Farrar, Straus, and Giroux.
- [Background] Bhana, D., & Pattman, R. (2009). Researching South African youth, gender and sexuality within the context of HIV/AIDS. Development, 52(1), 68-74.
- [Background] Reddy, S. P., Panday, S., Swart, D., Jinabhai, C. C., Amosun, S. L., James, S., Monyeki, K. D., Stevens, G., Morejele, N., Kambaran, N. S., Omardien, R. G., & Van den Borne, H.W. (2003). Umthenthe Uhlaba Usamila - The South African Youth Risk Behaviour Survey 2002. Cape Town, South Africa: South African Medical Research Council.
- [Background] South African Department of Health, Medical Research Council. (2007). South Africa Demographic and Health Survey 2003. Pretoria, South Africa: Department of Health.
- [Background] Coovadia H, Jewkes R, Barron P, Sanders D, McIntyre D. The health and health system of South Africa: historical roots of current public health challenges. Lancet. 2009 Sep 5;374(9692):817-34. doi: 10.1016/S0140-6736(09)60951-X. Epub 2009 Aug 24. PMID 19709728
- [Background] Parry CD. South Africa: alcohol today. Addiction. 2005 Apr;100(4):426-9. doi: 10.1111/j.1360-0443.2005.01015.x. PMID 15784051
- [Background] Scott-Sheldon LA, Carey MP, Carey KB, Cain D, Harel O, Mehlomakulu V, Mwaba K, Simbayi LC, Kalichman SC. Patterns of alcohol use and sexual behaviors among current drinkers in Cape Town, South Africa. Addict Behav. 2012 Apr;37(4):492-7. doi: 10.1016/j.addbeh.2012.01.002. Epub 2012 Jan 11. PMID 22273585
- [Background] Morojele NK, Kachieng'a MA, Mokoko E, Nkoko MA, Parry CD, Nkowane AM, Moshia KM, Saxena S. Alcohol use and sexual behaviour among risky drinkers and bar and shebeen patrons in Gauteng province, South Africa. Soc Sci Med. 2006 Jan;62(1):217-27. doi: 10.1016/j.socscimed.2005.05.031. Epub 2005 Jul 27. PMID 16054281
- [Background] Parry CD, Myers B, Morojele NK, Flisher AJ, Bhana A, Donson H, Pluddemann A. Trends in adolescent alcohol and other drug use: findings from three sentinel sites in South Africa (1997-2001). J Adolesc. 2004 Aug;27(4):429-40. doi: 10.1016/j.adolescence.2003.11.013. PMID 15288752
- [Background] Kalichman SC, Simbayi LC, Vermaak R, Jooste S, Cain D. HIV/AIDS risks among men and women who drink at informal alcohol serving establishments (Shebeens) in Cape Town, South Africa. Prev Sci. 2008 Mar;9(1):55-62. doi: 10.1007/s11121-008-0085-x. Epub 2008 Feb 9. PMID 18264762
- [Background] Parry, C. D. H., & Bennetts, A. L. (1998). Alcohol policy and public health in South Africa. Cape Town: Oxford University Press.
- [Background] Simbayi, L. C., Kalichman, S. C., Cain, D., Cherry, C., Henda, N., & Cloete, A. (2006). Methamphetamine use and sexual risks for HIV infection in Cape Town, South Africa. Journal of Substance Use, 11(4), 291-300.
- [Background] MRC Crime, Violence and Injury Lead Programme. (2003). A Profile of Fatal Injuries in South Africa. Fourth Annual Report of the National Injury Mortality Surveillance System. Pretoria: MRC.
- [Background] Jewkes R. Intimate partner violence: causes and prevention. Lancet. 2002 Apr 20;359(9315):1423-9. doi: 10.1016/S0140-6736(02)08357-5. PMID 11978358
- [Background] Jewkes RK, Dunkle K, Nduna M, Shai N. Intimate partner violence, relationship power inequity, and incidence of HIV infection in young women in South Africa: a cohort study. Lancet. 2010 Jul 3;376(9734):41-8. doi: 10.1016/S0140-6736(10)60548-X. PMID 20557928
- [Background] Michielsen K, Chersich MF, Luchters S, De Koker P, Van Rossem R, Temmerman M. Effectiveness of HIV prevention for youth in sub-Saharan Africa: systematic review and meta-analysis of randomized and nonrandomized trials. AIDS. 2010 May 15;24(8):1193-202. doi: 10.1097/QAD.0b013e3283384791. PMID 20375876
- [Background] UNAIDS. (2010). UNAIDS 2010 Report on the Global AIDS Epidemic. Retrieved from: http://www.unaids.org/globalreport/Global_report.htm
- [Background] Gupta GR, Parkhurst JO, Ogden JA, Aggleton P, Mahal A. Structural approaches to HIV prevention. Lancet. 2008 Aug 30;372(9640):764-75. doi: 10.1016/S0140-6736(08)60887-9. Epub 2008 Aug 5. PMID 18687460
- [Background] Dean HD, Fenton KA. Addressing social determinants of health in the prevention and control of HIV/AIDS, viral hepatitis, sexually transmitted infections, and tuberculosis. Public Health Rep. 2010 Jul-Aug;125 Suppl 4(Suppl 4):1-5. doi: 10.1177/00333549101250S401. No abstract available. PMID 20629250
- [Background] Harwood JM, Weiss RE, Comulada WS. Beyond the Primary Endpoint Paradigm: A Test of Intervention Effect in HIV Behavioral Intervention Trials with Numerous Correlated Outcomes. Prev Sci. 2017 Jul;18(5):526-533. doi: 10.1007/s11121-017-0788-y. PMID 28434056
- [Derived] Rotheram-Borus MJ, Tomlinson M, Stewart J, Skiti Z, Rabie S, Wang J, Almirol E, Vogel L, Christodoulou J, Weiss RE. Soccer and Vocational Training are Ineffective Delivery Strategies to Prevent HIV and Substance Abuse by Young, South African Men: A Cluster Randomized Controlled Trial. AIDS Behav. 2024 Dec;28(12):3929-3943. doi: 10.1007/s10461-024-04458-0. Epub 2024 Sep 11. PMID 39259241
- [Derived] Rabie S, Tomlinson M, Almirol E, Stewart J, Skiti Z, Weiss RE, Vogel L, Rotheram-Borus MJ. Utilizing Soccer for Delivery of HIV and Substance Use Prevention for Young South African Men: 6-Month Outcomes of a Cluster Randomized Controlled Trial. AIDS Behav. 2023 Mar;27(3):842-854. doi: 10.1007/s10461-022-03819-x. Epub 2022 Nov 15. PMID 36380117
- [Derived] Rabie S, Bantjes J, Gordon S, Almirol E, Stewart J, Tomlinson M, Rotheram-Borus MJ. Who can we reach and who can we keep? Predictors of intervention engagement and adherence in a cluster randomized controlled trial in South Africa. BMC Public Health. 2020 Feb 27;20(1):275. doi: 10.1186/s12889-020-8357-x. PMID 32106835
- [Derived] Christodoulou J, Stokes LR, Bantjes J, Tomlinson M, Stewart J, Rabie S, Gordon S, Mayekiso A, Rotheram-Borus MJ. Community context and individual factors associated with arrests among young men in a South African township. PLoS One. 2019 Jan 17;14(1):e0209073. doi: 10.1371/journal.pone.0209073. eCollection 2019. PMID 30653530
- [Derived] Rotheram-Borus MJ, Tomlinson M, Mayekiso A, Bantjes J, Harris DM, Stewart J, Weiss RE. Gender-specific HIV and substance abuse prevention strategies for South African men: study protocol for a randomized controlled trial. Trials. 2018 Aug 3;19(1):417. doi: 10.1186/s13063-018-2804-3. PMID 30075740